CLINICAL TRIAL: NCT01606969
Title: Randomized Controlled Trial to Comparison of Epinephrine-lidocaine Solution and Dexmedetomidine -Lidocaine Solution for the Effect on Hemodynamic Response Due to Scalp Infiltration in Patients Undergoing Craniotomy
Brief Title: Comparison of Epinephrine-lidocaine Solution and Dexmedetomidine -Lidocaine Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2012-0062
Record Dates: First submitted 2012-05-20; First posted 2012-05-28 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Craniotomy
Keywords: Dexmedetomidine; epinephrine; lidocaine; scalp infiltration; craniotomy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dex group (Experimental): dexmedetomidine-lidocaine solution,
  Interventions: Drug: scalp infiltration solution
- Control group (Active Comparator): epinephrine-lidocaine solution
  Interventions: Drug: scalp infiltration solution

INTERVENTIONS:
Drug: scalp infiltration solution — Dex group: Dexmedetomidine 2mcg/ml-containing 1% lidocaine scalp injection by neurosurgeon(dosage: according to incision length)
  Arms: Dex group
Drug: scalp infiltration solution — 1:100000 epinephrine-containing 1% lidocaine scalp injection by neurosurgeon(dosage: according to incision length)
  Arms: Control group

SUMMARY:
Scalp infiltration with Epinephrine- containing lidocaine solution is common method for craniotomy but it may result in transient but significant hypotension in patients undergoing neurosurgery. Dexmedetomidine, a potent alpha2 adrenoceptor agonist which dose-dependently reduces arterial blood pressure and heart rate, decreases the hemodynamic and catecholamine response, and dexmedetomidine has an effect of peripheral vasoconstriction thus it is thus theologically appropriate for reducing bleeding during scalp incision in craniotomy.

The aim of this study is to compare the effect of dexmedetomidine-lidocaine solution on hemodynamic response, scalp bleeding to epinephrine-lidocaine solution.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Aged between 20 and 70 year
* general anesthesia for craniotomy

Exclusion Criteria:

* Congestive heart failure, coronary artery occlusive disease
* Bradycardia < 50 BPM, 2nd degree < AV block
* Poorly controlled hypertension
* ß blocker medication
* Coagulopathy
* Pregnancy, nursing

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure | before and after scalp injection
  before scalp injection(T0), after scalp injection every half minute until five minutes(T0.5, T1, T1.5, T2, T2.5, T3, T3.5, T4, T4.5, T5), every minute(T6, T7, T8, T9, T10, T11, T12, T13, T14, T15)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea